CLINICAL TRIAL: NCT03425331
Title: Biomarkers of Response to Ipilimumab and Nivolumab as First-line Therapy for Metastatic Non-small Cell Lung Cancer (NSCLC): an Open-label, Single Arm Phase 2 Study
Brief Title: Biomarkers of Response to Ipilimumab and Nivolumab in First-line NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, competing studies, and lack of efficacy
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Biagio Ricciuti, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-566
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+Ipilimumab (Experimental): Nivolumab will be administered once every 2 weeks 1 mg/kg intravenously Ipilimumab will be administered once every 6 weeks 3 mg/kg intravenously
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab is a type of immunotherapy. Immunotherapy works by stimulating the body's own immune system to attack cancer cells
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab is a type of immunotherapy. Immunotherapy works by stimulating the body's own immune system to attack cancer cells
  Other Names: Opdivo

SUMMARY:
This research study is studying two immunotherapy drugs as a possible treatment for advanced non-small cell lung cancer (NSCLC).

The drugs involved in this study are:

* Ipilimumab
* Nivolumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of investigational drugs to learn whether the drugs work in treating a specific disease. "Investigational" means that the drugs are being studied.

The FDA (the U.S. Food and Drug Administration) has not approved ipilimumab for this specific disease but it has been approved for other uses, including for patients with advanced melanoma.

The FDA (the U.S. Food and Drug Administration) has approved nivolumab as a treatment option for this disease. However, nivolumab it is not approved in combination with ipilimumab to treat NSCLC.

Nivolumab and ipilimumab are both types of immunotherapy. Immunotherapy works by stimulating the body's own immune system to attack cancer cells. The combination of ipilimumab with nivolumab may or may not increase anti-cancer activity by further boosting the immune system.

In this research study, the investigators are investigating if the combination of ipilimumab and nivolumab is effective in treating advanced NSCLC. The investigators are also investigating whether there are certain DNA or protein markers in the blood or tumor tissue that may indicate whether the combination will work in future patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV NSCLC, with no prior systemic anti-cancer therapy of any kind (including EGFR and ALK inhibitors). Prior definitive chemoradiation for locally advanced disease is permitted as long as the last administration of chemotherapy or radiation (whichever was given last) occurred at least 6 months prior to enrollment. Prior adjuvant or neoadjuvant chemotherapy for early stage lung cancer is permitted if completed at least 6 months prior to initiating study treatment.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Age ≥ 18 years.
* ECOG performance status ≤ 1 (see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN, OR
  * AST(SGOT)/ALT(SGPT) ≤ 5 × institutional ULN if liver metastases are present
  * Serum creatinine ≤ 1.5 × institutional ULN, OR
  * Creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with serum creatinine levels above 1.5 × institutional ULN.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must have a tumor tissue sample available (formalin-fixed paraffin embedded [FFPE] tissue block or unstained slides); may be newly obtained or obtained within 6 months prior to enrollment (without systemic therapy given after the sample was obtained). Participants without sufficient archival tissue may be enrolled following successful completion of the pre-treatment tumor tissue biopsy. Tissue must be a core needle biopsy, excisional, or incisional biopsy. Fine needle aspirates (FNA) or malignant effusions are not adequate. Bone biopsies without a soft tissue component are not adequate.
* The effects of nivolumab and ipilimumab on the developing human fetus are unknown. For this reason, women of childbearing potential (WOCBP) must agree to follow instructions for acceptable contraception from the time of signing consent, and for 23 weeks after their last dose of protocol-indicated treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol who are not azoospermic who are sexually active with WOCBP must agree to follow instructions for acceptable contraception from the time of signing consent, and for 31 weeks after their last dose of protocol-indicated treatment.
* Participants must be able and willing to undergo a pre-treatment tumor tissue biopsy. Participants must also be willing to undergo an on-treatment tumor tissue biopsy if clinically feasible.

Exclusion Criteria:

* Participants with known EGFR mutations or ALK rearrangements. All subjects must have been tested for EGFR mutation and ALK rearrangement prior to study entry, unless they are known to have a KRAS mutation.
* Participants who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Participants who received prior non-CNS directed palliative radiation therapy within 7 days of the date of study entry.
* Participants who are receiving any other investigational agents.
* Participants with known untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Subjects are eligible if CNS metastases are adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to study entry. Subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent) for at least 2 weeks prior to first study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ipilimumab or nivolumab.
* Participants with previous malignancies are excluded unless a complete remission was achieved at least 2 years prior to first treatment and no additional therapy is required or anticipated to be required during the study period as judged by the treating investigator. Exceptions include non-melanoma skin cancers, and in situ cancers of any type (e.g. bladder, gastric, colon, cervical/dysplasia, melanoma, or breast carcinoma in situ).
* Participants with any other active malignancy requiring concurrent intervention.
* Participants with an active, known, or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with corticosteroids of > 10 mg daily prednisone (or equivalent), or subjects requiring other immunosuppressive medications within 14 days of first treatment. Inhaled, topical, ophthalmologic, local steroid injections, and adrenal replacement steroid > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
* Participants with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity in the opinion of the treating investigator.
* Participants with a known history of testing positive for human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS).
* Participants with known positive test for hepatitis B or C indicating acute or chronic infection.
* Participants with ≥ Grade 2 peripheral neuropathy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ipilimumab and nivolumab are both agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ipilimumab or nivolumab, breastfeeding should be discontinued if the mother is treated with ipilimumab or nivolumab. A negative serum pregnancy test is required prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2021-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Awad, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 04/2018 to 11/2018.
Groups:
- Nivolumab+Ipilimumab: Nivolumab will be administered once every 2 weeks at a dosage of 3 mg/kg intravenously and Ipilimumab will be administered once every 6 weeks at a dosage of 1 mg/kg intravenously
Period: Overall Study
Arm/Group | Nivolumab+Ipilimumab
Started | 5
Completed | 0
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Groups:
- Nivolumab+Ipilimumab: Nivolumab will be administered once every 2 weeks at a dosage of 3 mg/kg intravenously, and Ipilimumab will be administered once every 6 weeks at a dosage of 1 mg/kg intravenously
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.80 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Response
Description: Best response on treatment is based on RECISTv1.1 criteria: Complete Response (CR) is complete disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Both require confirmation no fewer than 4 weeks apart. Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, and the sum must also demonstrate an absolute increase of at least 5 mm since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Stable Disease (SD) is defined as any condition not meeting the above criteria.
Time Frame: Disease was evaluated radiologically at baseline and then every 6 weeks for the first 6 cycles of therapy. Median treatment duration for this study cohort is 8.05 months with range (2.76 months - 15.90 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 5
Participants
  Partial Response | 3
  Stable Disease | 2

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the duration between registration and documented disease progression (PD) defined per RECIST 1.1 criteria or death, or is censored at time of last disease assessment.
Time Frame: Disease was evaluated at baseline and then every 6 weeks for the first 6 cycles of therapy and in long-term follow-up every 3 months. Median follow-up for survival is of 15.97 months with range (4.00 months - 20.63 months).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 5
months | 6.90 [4.01 to NA] — There are only 3 events, therefore the upper limit of the 90% CI is not finite.

3. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Median follow-up for survival is of 15.97 months with range (4.00 months - 20.63 months).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 5
months | 15.97 [15.31 to NA] — There are only 3 events, therefore the upper limit of the 90% CI is not finite.

4. Secondary Outcome: Median Duration of Response (DOR)
Description: DOR, estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per RECISTv1.1, until the first date that recurrent or progressive disease is objectively documented. Patients without PD are censored at the date of last disease assessment.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 5
months | 4.11 [2.74 to 8.39]

5. Secondary Outcome: Incidence of Grade 4-5 Treatment-related Toxicity Rate
Description: All grade 4-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.
Time Frame: AE evaluated on day 1, 15, 29 each cycle. The median of treatment duration is 8.05 months with range (2.76 months - 15.90 months).
Measure: Number; unit: proportion of participants
Arm/Group | Nivolumab+Ipilimumab
Number analyzed (Participants) | 5
proportion of participants | 0.2

ADVERSE EVENTS:
Time Frame: AE evaluated on day 1, 15, 29 each cycle on treatment. The median of the observation period for all-cause mortality is 15.97 months with range (4.00 months - 20.63 months). The median of observation time for AE is 8.05 months with range (2.76 months - 15.90 months).
Description: A SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event, requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event, suspected transmission of an infectious agent via the study drug is an SAE
Arm/Group | Nivolumab+Ipilimumab
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Ipilimumab (N=5)
Adrenal insufficiency (Endocrine disorders) | 1
Fever (General disorders and administration site conditions) | 1
Lung infection (Infections and infestations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Ipilimumab (N=5)
Anemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders and administration site conditions) | 2
Fatigue (General disorders and administration site conditions) | 3
Fever (General disorders and administration site conditions) | 1
Non-cardiac chest pain (General disorders and administration site conditions) | 3
Pain (General disorders and administration site conditions) | 1
Bronchial infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 1
Lipase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Serum amylase increased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03425331/Prot_SAP_000.pdf